CLINICAL TRIAL: NCT07133932
Title: Transcutaneous Electrical Phrenic Nerve Stimulation for Reducing Mechanical Ventilation Duration in Acute Cerebral Infarction: A Multicenter Randomized Controlled Trial
Brief Title: Phrenic Nerve Stimulation for Reducing Ventilation Duration in Acute Cerebral Infarction: A Multicenter Randomized Controlled Trial
Acronym: EDP-VENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-161-002
Record Dates: First submitted 2025-07-21; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Infarction; Mechanical Ventilation; Acute Cerebrovascular Accident; Adult
MeSH Terms: conditions — Cerebral Infarction; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Transcutaneous electrical phrenic nerve stimulation for 14 days
  Interventions: Device: Transcutaneous electrical phrenic nerve stimulation
- Control group (Sham Comparator): Sham stimulation for 14 days
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Transcutaneous electrical phrenic nerve stimulation — Non-invasive transcutaneous electrical phrenic nerve stimulation which can cause explicit contraction of the diaphragm, and the stimulation current may be set to 5-30mA depending on the participant's condition.
  Arms: Intervention group
Device: Sham (No Treatment) — The stimulation current is set to 0.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if non-invasive phrenic nerve stimulation works in adult acute cerebral infarction participants undergoing mechanical ventilation. It will also learn about the safety of non-invasive phrenic nerve stimulation. The main questions it aims to answer are：

1. Can non-invasive phrenic nerve stimulation shorten the duration of ventilator use and improve long-term prognosis?
2. What medical problems do participants have when taking non-invasive phrenic nerve stimulation? Researchers will compare non-invasive phrenic nerve stimulation to a sham stimulation to see if non-invasive phrenic nerve stimulation works.

Participants will:

1. Receive 14 days of non-invasive phrenic nerve stimulation or sham stimulation
2. Visit the clinic or call for follow-up at 90 days of onset

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* no gender restrictions
* patient diagnosed with acute cerebral infarction (within 30 days of onset) through cranial CT or MRI
* duration of mechanical ventilation ≥ 24 hours
* patient or their legal guardian agrees to participate in the study and signs an informed consent form

Exclusion Criteria:

* there are other significant conditions that affect diaphragm function, such as severe malnutrition, irreversible respiratory pump failure caused by medullary or cervical cord injury, and irreversible damage to the phrenic nerve
* significant agitation cannot be combined with transcutaneous electrical phrenic nerve stimulation
* severe skin damage or infection at the electrode placement site
* previous presence of severe lung disease (such as severe COPD, interstitial lung disease, pulmonary embolism, etc.), severe heart failure (NYHA Class IV)
* sepsis or shock requiring high-dose vasopressors
* the terminal state of the disease or expected survival period does not exceed 7 days
* pacemaker implantation
* pregnant or lactating women
* patients whose family members express their willingness to withdraw for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mechanical ventilation duration | Successfully weaned from ventilater for 48 hours
  The total duration of mechanical ventilation, which is the time difference between starting mechanical ventilation and successfully weaning.

SECONDARY OUTCOMES:
Successful weaning rate | Successfully weaned from ventilater for 48 hours
mRS at 90 days | 90 days of symptom onset

OTHER OUTCOMES:
Tracheostomy rate | Through ICU discharge, up to 90 days
In-hospital mortality | Through ICU discharge, up to 90 days
Mortality at 90 days | 90 days of symptom onset
ICU length of stay | Through ICU discharge, up to 90 days
ICU cost | Through ICU discharge, up to 90 days
Quality of Life (EQ-5D-5L score) at 90 days | 90 days of symptom onset
Incidence rate of ventilator-associated pneumonia | Through ICU discharge, up to 90 days
Incidence rate of ventilator-induced diaphragmatic dysfunction | Through ICU discharge, up to 90 days
Number of participants with electrode patch-associated skin injury | Day 14

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Hospital of Heibei Medical University, Shijiazhuang, Hebei
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Hui Min Hospital, Beijing
  - Sanbo Brain Hospital, Capital Medical University, Beijing
  - Dongzhimen Hospital Beijing University of Chinese Medicine, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - The First Hospital of Fangshan District, Beijing
  - Beijing Daxing District People's Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Yes
After the research is completed and the results are published, the project leader can be contacted to obtain the original data.
Supporting Information: Study Protocol, SAP, CSR